CLINICAL TRIAL: NCT01561105
Title: This Was a Five-year Seven-site Trial to Study the Cost-effectiveness of a Population Based Disease Management Program for Late Life Depression in Primary Care.
Brief Title: Improving Depression Care for Elders: Coordinating Center
Acronym: IMPACT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: The John A. Hartford Foundation (Other); California HealthCare Foundation (Other); Hogg Foundation (Unknown); Robert Wood Johnson Foundation (Other)
Responsible Party: Principal Investigator, Jurgen Unutzer, MD, MPH, Professor and Vice-Chair of Psychiatry, Psychiatry and Behavioral Sciences, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: JAHF 98297
Record Dates: First submitted 2012-03-20; First posted 2012-03-22 (Estimated); Last update posted 2012-03-28 (Estimated); Status verified 2012-03

CONDITIONS: Major Depression; Dysthymic Disorder; Both Major Depression and Dysthymic Disorder
MeSH Terms: conditions — Depressive Disorder, Major; Dysthymic Disorder

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- IMPACT (Experimental)
  Interventions: Other: IMPACT
- Care as Usual (No Intervention): Patients received all depression care available to them as part of care as usual in the participating primary care clinics.

INTERVENTIONS:
Other: IMPACT — IMPACT is a collaborative care management program for late-life depression
  Other Names: Improving Mood-Promoting Access to Collaborative Treatment
  Arms: IMPACT

SUMMARY:
Purpose: To determine the effectiveness of the Improving Mood-Promoting Access to Collaborative Treatment(IMPACT) collaborative care management program for late-life depression.

DETAILED DESCRIPTION:
This study tested an organized method of delivering care for late life depression in primary care. Specifically, the investigators evaluated the effectiveness of this intervention as compared to 'care as usual'. The investigators studied the effect of the intervention on clinical outcomes such as depressive symptoms, functional status, health related quality of life. They also determined the cost-effectiveness of the intervention compared to care as usual.

ELIGIBILITY:
Inclusion Criteria:

* Major depression or dysthymia as diagnosed by a structured diagnostic interview.
* Patient plans to receive primary care at the study clinic for the next year.

Exclusion Criteria:

* Age under 60.
* Current symptoms or history of psychosis or mania as determined by structured diagnostic interview.
* Cognitive impairment as defined by a score less than 23 on a Mini Mental Status Examination.
* Terminal illness - defined as having a life expectancy of less than 6 months.
* Active alcohol abuse as determined by a screening interview.
* High suicide risk as determined by current plan for suicide or a history of more than 3 prior suicide attempts in the past 10 years.

Min Age: 60 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 1801 (Actual)
Dates: Start 1999-01; Primary Completion 2004-06 (Actual); Study Completion 2004-06 (Actual)

PRIMARY OUTCOMES:
Severity of depression symptoms
  Severity measured by the 21-item Hopkins Symptom Checklist.

SECONDARY OUTCOMES:
Functioning
  measured by the Sheehan Health-Related Functioning Index

CONTACTS AND LOCATIONS:
Overall Officials: Jurgen Unutzer, MD, MPH, Principal Investigator — University of Washington

REFERENCES:
- [Result] Unutzer J, Katon W, Callahan CM, Williams JW Jr, Hunkeler E, Harpole L, Hoffing M, Della Penna RD, Noel PH, Lin EH, Arean PA, Hegel MT, Tang L, Belin TR, Oishi S, Langston C; IMPACT Investigators. Improving Mood-Promoting Access to Collaborative Treatment. Collaborative care management of late-life depression in the primary care setting: a randomized controlled trial. JAMA. 2002 Dec 11;288(22):2836-45. doi: 10.1001/jama.288.22.2836. PMID 12472325
- [Derived] Stewart JC, Perkins AJ, Callahan CM. Effect of collaborative care for depression on risk of cardiovascular events: data from the IMPACT randomized controlled trial. Psychosom Med. 2014 Jan;76(1):29-37. doi: 10.1097/PSY.0000000000000022. Epub 2013 Dec 23. PMID 24367124